CLINICAL TRIAL: NCT03531333
Title: Intraoperative Ultrasound Guidance and Extent of Resection in High Grade Glioma Surgery: a Randomised, Controlled Trial.
Brief Title: Intraoperative Ultrasound Guided Glioma Surgery; a Randomised, Controlled Trial.
Acronym: US-GLIOMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Stichting Coolsingel (Unknown)
Responsible Party: Principal Investigator, A.J.P.E. VIncent, neurosurgeon, principal investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEC-2015-46
Record Dates: First submitted 2017-11-02; First posted 2018-05-21 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Glioma
Keywords: Glioma, intraoperative ultrasound, gross total resection, quality of life
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: The US-GLIOMA study is a randomized controlled trial with blinded primary outcome measure.
  The study consists of two treatment arms: non-ultrasound guided glioma resection (conventional treatment) versus ultrasound guided glioma resection (intervention) .
Who Masked: Outcomes Assessor
Masking Description: Gross total resection (yes/no) on post-operative T1 postcontrast MRI scans will be evaluated by a neuroradiologist who is blinded for the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound (Experimental): ultrasound navigation guided surgery.
  Interventions: Procedure: ultrasound guided surgery.
- Non-ultrasound (No Intervention): standard surgery without ultrasound guidance.

INTERVENTIONS:
Procedure: ultrasound guided surgery. — during surgery, the neurosurgeon will acquire ultrasound guided images (fused with the standard neuronavigation system) to evaluate the progress of tumor resection.
  Arms: Ultrasound

SUMMARY:
The main goal of high grade glioma (HGG) surgery is to achieve gross total resection (GTR) without causing new neurological deficits1-8. Intraoperative navigated high resolution ultrasound (US) is a promising new tool to acquire real-time intraoperative images to localize and to resect gliomas9-12. The aim of this study was to investigate whether intraoperative guided surgery leads to a higher rate of GTR, when compared with standard non-ultrasound guided surgery.

DETAILED DESCRIPTION:
Study design:

The US-GLIOMA study is a randomized controlled trial with blinded primary outcome measure.

Study population:

Fifty patients with newly diagnosed contrast enhancing presumed high grade glioma on first MRI scan.

Intervention:

The study consists of two treatment arms: non-ultrasound guided glioma resection (conventional treatment) versus ultrasound guided glioma resection (intervention) .

Main study parameters/endpoints:

* Gross total resection (yes/no)
* Extent of resection (%)
* Neurological outcome (Karnofsky Performance Status)
* Quality of Life (EORTC QLQ-C30 and QLQ-BN20 quality of life questionnaire)
* Surgery associated neurological deficits (National Institutes of Health Stroke Scale)
* Adverse events (classified according to the US National Cancer Institute common toxicity criteria version 4.0)
* Survival time (days)

ELIGIBILITY:
Inclusion Criteria:

* Individuals of 18 years or older
* Newly diagnosed, untreated, contrast enhancing presumed high-grade glioma
* KPS ≥ 60
* Preoperative intention to perform gross-total resection of the enhancing tumor
* Written informed consent conform ICH-GCP

Exclusion Criteria:

* Tumours crossing the midline basal ganglia, cerebellum, or brain stem prohibiting gross total resection
* Multifocal contrast enhancing lesions
* Pre-existing neurological deficit (e.g. aphasia, hemiparesis) due to neurological diseases (e.g. stroke)
* Inability to give consent because of dysphasia or language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Gross total resection (Yes or No) | within 48 hours after surgery
  Gross-total resection (yes vs. no): No residual contrast enhancement on post-operative MRI scans; 100% of all contrast enhancing tumor has been resected when compared to initial enhancing tumor on pre-operative MRI scans.

SECONDARY OUTCOMES:
Extent of resection (%) | within 48 hours after surgery
  as a continous variable The extent of resection (%) is a secondary outcome measurement defined as the residual tumor volumes on post-operative MRI studies compared to the operative tumor volume.
Neurological outcome (Karnofsky Performance status) | within 1 week after surgery
  Karnofsky Performance status
Quality of Life (QLQ C30 questionnaires) | 1, 3 and 6 months after surgery
  QLQ C30 questionnaires
  A brain tumor specific quality of life measurement tool
Quality of Life (QLQ BN20 questionnaires) | 1, 3 and 6 months after surgery
  QLQ BN20 questionnaires
  A brain tumor specific quality of life measurement tool
Surgery associated neurological deficits (National Institutes of Health Stroke Scale) | 1 month after surgery
  National Institutes of Health Stroke Scale
  0 No stroke symptoms 1-4 Minor stroke 5-15 Moderate stroke 16-20 Moderate to severe stroke 21-42 Severe stroke
  NIHSS is a tool used by healthcare providers to objectively quantify the impairment caused typically by a stroke, however it is also used for tumor studies to assess functioning on the level of speech, motor and sensory functions.
Survival (time in days) | status will be checked 15 months after surgery
  time measured from surgery until death in days.
  This study has a follow up of 6 months. However, when patients are alive at months after surgery, we will contact the general practictioner of the patient 15 months after the trial to obtain survival data.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Incekara F, Smits M, Dirven L, Bos EM, Balvers RK, Haitsma IK, Schouten JW, Vincent AJPE. Intraoperative B-Mode Ultrasound Guided Surgery and the Extent of Glioblastoma Resection: A Randomized Controlled Trial. Front Oncol. 2021 May 19;11:649797. doi: 10.3389/fonc.2021.649797. eCollection 2021. PMID 34094939